CLINICAL TRIAL: NCT04071522
Title: Cross-Cultural Adaptation and Validation of the Back Beliefs Questionnaire to the Turkish Language
Brief Title: Validation of the Back Beliefs Questionnaire to the Turkish
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: 050.05.04.05.01
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Low Back Pain
Keywords: low back pain; turkish language; pain beliefs; validity
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LBP: 110 literate Turkish speaking patients suffering from low back pain (LBP) for over 3 months, within the age range 18-65 were included in the study.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The Back Beliefs Questionnaire (BBQ) developed by Symonds et al. in 1996 is used to measure patient's attitudes and beliefs towards recovery and return-to-work; and expectations regarding the negative circumstances that could be created as a result of low back pain (LBP).The aim of this study was the translation to Turkish language, cross-cultural adaptation and assessment of reliability&validity of BBQ for the patients suffering from chronic LBP.

DETAILED DESCRIPTION:
Back Beliefs Questionnaire was translated and culturally adapted into Turkish regarding to the published guidelines. This observational cross-sectional study was performed with 110 chronic low back pain patients. All participants were asked to complete Back Beliefs Questionnaire and also fill the socio-demographic data form and evaluation tools (Numeric rating scale-pain, Oswestry Disability Index, Fear Avoidance Beliefs Questionnaire, Hospital Anxiety and Depression Scale). Internal consistency was evaluated with Cronbach's alfa coefficient. Intraclass correlation coefficient was used to assess test-retest reliability. Structural validity was assessed by correlations with other tools.

Back Beliefs Questionnaire had a good internal consistency (Cronbach alfa= 0.79) and an excellent test-retest reliability (Intraclass correlation coefficient = 0.84). A moderate correlation was determined between Back Beliefs Questionnaire and Fear Avoidance Beliefs Questionnaire. Correlations with Numeric rating scale-pain, Oswestry Disability Index, Hospital Anxiety and Depression Scale were fair.

Turkish version of Back Beliefs Questionnaire is a valid and reliable questionnaire that can be used to evaluate beliefs about pain in patients with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Turkish speaking
* Suffering from low back pain during activity for over 3 months

Exclusion Criteria:

* pregnancy
* malignancy
* infections
* fractures
* inflammatory diseases
* cognitive impairments that might create a problem in comprehending and filling the survey

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who consulted to our Physical Medicine and Rehabilitation clinic during the period between June 2018 and April 2018; and volunteered to participate in this study were evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Back Beliefs Questionnaire | 10 minutes
  BBQ was designed to evaluate patients' LBP and their expectations regarding the negative outcomes that might be inflicted on their future; and their attitude towards return-to-work.BBQ consists of 14 items to be filled in by patients. Nine of which are used to evaluate inevitability (1st, 2nd, 3rd, 6th, 8th, 10th, 12th, 13th, 14th) and the other 5 are distractors (4th, 5th, 7th, 9th, 11th). All items are evaluated on a 5-point-Likert Scale that referred to "1-Definitely Disagree" and "5-Definitely Agree". Scoring is calculated over the expressions included in the inevitability measure by reversing the numerical values which are appointed by the participants. The resulting score is between 9 and 45. Lower scores supports the more incompatible and pessimistic beliefs.
Numeric Rating Scale-Pain | 2 minutes
  Numeric Rating Scale-Pain is a scale with good sensitivity that quantitatively evaluates the pain intensity, which is easily comparable to other pain scales. The patient defines pain level within a range of 1 to 10. 1 point represents the minumum pain level, while 10 indicates the most severe pain.
Oswestry Disability Index | 5 minutes
  Oswestry Disability Index is a scale that assesses the functional disability level associated with LBP. It consists of 10 items that each have 6 options, which are scored between 0-5. The patient's total score is divided by the maximum possible score and multiplied by 100; and a percentage score is thus attained. The resulting score is between 0 and 100. As the total score increases, the level of functional disability also increases
Fear Avoidance Beliefs Questionnaire | 3 minutes
  Fear Avoidance Beliefs Questionnaire evaluates the physical activity and work related beliefs of fear and avoidance that arise in patients with LBP. It consists of two subscales (physical activity and work) and 16 questions in total.The patient rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs.
Hospital Anxiety and Depression Scale | 3 minutes
  The Hospital Anxiety and Depression Scale is a frequently used self-rating scale developed to assess psychological distress in non-psychiatric patients. The questionnaire comprises seven questions for anxiety and seven questions for depression. HADS scores were interpreted as follows for each subscale: mild=8-10, modarate=11-14, severe=15-21.

CONTACTS AND LOCATIONS:
Locations (1):
- BezmialemVU, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will not be shared.

REFERENCES:
- [Background] Freburger JK, Holmes GM, Agans RP, Jackman AM, Darter JD, Wallace AS, Castel LD, Kalsbeek WD, Carey TS. The rising prevalence of chronic low back pain. Arch Intern Med. 2009 Feb 9;169(3):251-8. doi: 10.1001/archinternmed.2008.543. PMID 19204216
- [Background] Meucci RD, Fassa AG, Paniz VM, Silva MC, Wegman DH. Increase of chronic low back pain prevalence in a medium-sized city of southern Brazil. BMC Musculoskelet Disord. 2013 May 1;14:155. doi: 10.1186/1471-2474-14-155. PMID 23634830
- [Background] Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gosselin R, Grainger R, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Ma J, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2163-96. doi: 10.1016/S0140-6736(12)61729-2. PMID 23245607
- [Background] Waddell G, Newton M, Henderson I, Somerville D, Main CJ. A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability. Pain. 1993 Feb;52(2):157-168. doi: 10.1016/0304-3959(93)90127-B. PMID 8455963
- [Background] Linton SJ, Buer N, Vlaeyen J, Hellsing AL. Are fear-avoidance beliefs related to the inception of an episode of back pain? A prospective study. Psychol Health. 2000 Nov;14(6):1051-9. doi: 10.1080/08870440008407366. PMID 22175261
- [Background] Burton AK, Waddell G, Tillotson KM, Summerton N. Information and advice to patients with back pain can have a positive effect. A randomized controlled trial of a novel educational booklet in primary care. Spine (Phila Pa 1976). 1999 Dec 1;24(23):2484-91. doi: 10.1097/00007632-199912010-00010. PMID 10626311
- [Background] Symonds TL, Burton AK, Tillotson KM, Main CJ. Do attitudes and beliefs influence work loss due to low back trouble? Occup Med (Lond). 1996 Feb;46(1):25-32. doi: 10.1093/occmed/46.1.25. PMID 8672790
- [Background] Ferreira ML, Machado G, Latimer J, Maher C, Ferreira PH, Smeets RJ. Factors defining care-seeking in low back pain--a meta-analysis of population based surveys. Eur J Pain. 2010 Aug;14(7):747.e1-7. doi: 10.1016/j.ejpain.2009.11.005. Epub 2009 Dec 24. PMID 20036168
- [Background] Steenstra IA, Koopman FS, Knol DL, Kat E, Bongers PM, de Vet HC, van Mechelen W. Prognostic factors for duration of sick leave due to low-back pain in dutch health care professionals. J Occup Rehabil. 2005 Dec;15(4):591-605. doi: 10.1007/s10926-005-8037-9. PMID 16254758
- [Background] Alexopoulos EC, Konstantinou EC, Bakoyannis G, Tanagra D, Burdorf A. Risk factors for sickness absence due to low back pain and prognostic factors for return to work in a cohort of shipyard workers. Eur Spine J. 2008 Sep;17(9):1185-92. doi: 10.1007/s00586-008-0711-0. Epub 2008 Jul 23. PMID 18649089
- [Background] Haahr JP, Frost P, Andersen JH. Predictors of health related job loss: a two-year follow-up study in a general working population. J Occup Rehabil. 2007 Dec;17(4):581-92. doi: 10.1007/s10926-007-9106-z. Epub 2007 Oct 24. PMID 17957450
- [Background] Frazier LM, Carey TS, Lyles MF, McGaghie WC. Lengthy bed rest prescribed for acute low back pain: experience at three general medicine walk-in clinics. South Med J. 1991 May;84(5):603-6. PMID 1827930
- [Background] Elfering A, Muller U, Rolli Salathe C, Tamcan O, Mannion AF. Pessimistic back beliefs and lack of exercise: a longitudinal risk study in relation to shoulder, neck, and back pain. Psychol Health Med. 2015;20(7):767-80. doi: 10.1080/13548506.2015.1017824. Epub 2015 Mar 2. PMID 25726859
- [Background] Godges JJ, Anger MA, Zimmerman G, Delitto A. Effects of education on return-to-work status for people with fear-avoidance beliefs and acute low back pain. Phys Ther. 2008 Feb;88(2):231-9. doi: 10.2522/ptj.20050121. Epub 2007 Dec 4. PMID 18056753
- [Background] Chen G, Tan BK, Jia HL, O'Sullivan P, Burnett A. Questionnaires to examine Back Pain Beliefs held by health care professionals: a psychometric evaluation of Simplified Chinese versions. Spine (Phila Pa 1976). 2011 Aug 15;36(18):1505-11. doi: 10.1097/BRS.0b013e3181f49eec. PMID 21240047
- [Background] Alamrani S, Alsobayel H, Alnahdi AH, Moloney N, Mackey M. Cross-Cultural Adaptation and Validation of the Back Beliefs Questionnaire to the Arabic Language. Spine (Phila Pa 1976). 2016 Jun;41(11):E681-E686. doi: 10.1097/BRS.0000000000001341. PMID 27244114
- [Background] Dupeyron A, Lanhers C, Bastide S, Alonso S, Toulotte M, Jourdan C, Coudeyre E. The Back Belief Questionnaire is efficient to assess false beliefs and related fear in low back pain populations: A transcultural adaptation and validation study. PLoS One. 2017 Dec 6;12(12):e0186753. doi: 10.1371/journal.pone.0186753. eCollection 2017. PMID 29211745
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Background] Fairbank JC. Oswestry disability index. J Neurosurg Spine. 2014 Feb;20(2):239-41. doi: 10.3171/2013.7.SPINE13288. Epub 2013 Nov 22. No abstract available. PMID 24266676
- [Background] Roland M, Fairbank J. The Roland-Morris Disability Questionnaire and the Oswestry Disability Questionnaire. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3115-24. doi: 10.1097/00007632-200012150-00006. No abstract available. PMID 11124727